CLINICAL TRIAL: NCT00303394
Title: Phase 2 Study of IL-1Ra in Patients With Type 2 Diabetes
Brief Title: Treatment of Patients With Type 2 Diabetes With an Interleukin-1 Antagonist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: EK-1000-ZH
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes, IL-1, inflammation, glucotoxicity, insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Insulin Resistance | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Drug: IL-1Ra

SUMMARY:
Aim: To investigate the therapeutic potential of IL-1Ra in type 2 diabetes.

Rationale: Since the major defect leading to a decrease in b-cell mass in type 2 diabetes is increased apoptosis, therapeutic approaches designed to arrest apoptosis could be a significant new development in its management. This approach might actually reverse the disease to a degree rather than just palliate glycemia. Based on current thinking, treatment with IL-1Ra appears as a promising approach. The prospected effect is blocking of the IL-1b-mediated glucotoxicity and thereby to prevent the decline in b-cell mass, together with a rapid restoration of b-cell function. FDA approval for IL-1Ra in the treatment of rheumatoid arthritis occurred based on a favourable tolerability profile.

DETAILED DESCRIPTION:
Methodology: This will be a two-centre (University Hospital, Zurich, Switzerland and Steno Diabetes Center, Gentofte, Denmark) study. 72 patients will be randomised according to a double-blind, placebo-controlled protocol in which half of the patients are treated with IL-1Ra, the other half with saline. The treatment period will last 13 weeks. This time-period should be sufficient for reversal of functional glucotoxicity and feasible in terms of patient compliance. Whether 13 weeks of treatment will be sufficient to make significant changes in b-cell mass in unpredictable. However, blocking b-cell apoptosis, while new islet formation and b-cell replication are normal, may initiate enlargement of b-cell mass, which may progress beyond the treatment period. Patient evaluation will be performed at start and after 4, 13, 26, 39 and 52 weeks. Following 13 weeks, patients with a fasting plasma glucose levels > 8 mM or with a glycosylated hemoglobin level (HbA1c) > 8% will be treated with insulin. Insulin treatment will not be initiated earlier to avoid interference with possible effects of insulin on primary outcome in the period where the largest effect of IL-1Ra are expected. To assess effects of IL-1Ra on insulin sensitivity, a subset of 40 patients (20 IL-1Ra- and 20 placebo-treated) will undergo an euglycemic-hyperinsulinemic clamp as well as a muscle and fat biopsy at start and after the end of treatment (13 weeks). The Ethics Committee of both centres have already approved the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age >20
* Diabetes mellitus Type 2 (American Diabetes Association criteria) of at least 3 months duration
* HbA1c >7.5%
* Body-mass index (BMI) > 27

Exclusion Criteria:

* Positive GAD 65 or IA-2 antibodies at inclusion.
* HbA1c >12%, polyuria and thirst (exclusion of severely decompensated patients)
* C-peptide < 400pmol/l (basal )
* Established anti-inflammatory therapy (includiung cortisone, NSAID, Cox-2-inhibitor). Low dose aspirin (£ 100mg) will be tolerated.
* CRP >30 mg/dl, fever, current treatment with antibiotics, or chronic granulomatous infections (e.g. tuberculosis) in the history or on a screening chest X-ray.
* Neutropenia or anemia (leucocyte count < 2.0x109 /l, hemoglobin <11g/dl for ma les or <10g/dl for females)
* Pregnancy or breast-feeding. When appropriate (fertile women),anticonception for at last 3 month prior inclusion will be required.
* Severe liver or renal disease ( AST or ALT>3 times the upper limit of normal laboratory range, serum creatinine >130mM)
* Ongoing malignant neoplasm
* Use of any investigational drug within 30 days of enrollment into the study or within 5 half-lives of the investigational drug (whichever is longer)
* Immunosuppressive treatment or immunodeficient diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2004-04; Study Completion 2006-03

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
Insulin requirement
Stimulated C peptide and insulin
Fasting plasma glucose (FPG)
Serum cytokine levels, CRP
Insulin secretion and Insulin-sensitivity index derived from an OGTT with insulin and glucose measurements.
In a subgroup of patients, insulin-sensitivity assessed by clamp techniques
Insulin signaling- and cytokine- gene expression profiles derived from muscle and fat biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, MD, Study Chair — University of Zurich
Locations (2):
- Steno Diabetes Center, Gentofte Municipality, Copenhagen, Denmark
- University Hospital of Zurich, Division of Endocrinology and Diabetes, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] de Baat A, Trinh B, Ellingsgaard H, Donath MY. Physiological role of cytokines in the regulation of mammalian metabolism. Trends Immunol. 2023 Aug;44(8):613-627. doi: 10.1016/j.it.2023.06.002. Epub 2023 Jul 7. PMID 37423882
- [Derived] Larsen CM, Faulenbach M, Vaag A, Volund A, Ehses JA, Seifert B, Mandrup-Poulsen T, Donath MY. Interleukin-1-receptor antagonist in type 2 diabetes mellitus. N Engl J Med. 2007 Apr 12;356(15):1517-26. doi: 10.1056/NEJMoa065213. PMID 17429083